CLINICAL TRIAL: NCT02315196
Title: A Phase 2 Trial of Liposomal Doxorubicin and Carboplatin in Patients With ER, PR, HER2 Negative Breast Cancer (TNBC)
Brief Title: Pegylated Liposomal Doxorubicin Hydrochloride and Carboplatin Followed by Surgery and Paclitaxel in Treating Patients With Triple Negative Stage II-III Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Principal Investigator, Deborah Toppmeyer, MD, Professor of Medicine, Rutgers Cancer Institute of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 041401; NCI-2014-02029 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro20140000477041401 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2014-10-28; First posted 2014-12-11 (Estimated); Results first posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Estrogen Receptor-negative Breast Cancer; HER2-negative Breast Cancer; Progesterone Receptor-negative Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Triple-negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — liposomal doxorubicin; Epirubicin; Carboplatin; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (doxil, carboplatin, surgery, paclitaxel) (Experimental): NEOADJUVANT: Patients receive pegylated liposomal doxorubicin hydrochloride* IV over 90 minutes and carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  ADJUVANT: Patients undergo definitive surgery at the discretion of the treating physician. Patients then receive paclitaxel IV over 60 minutes once weekly for 12 weeks in the absence of disease progression or unacceptable toxicity.
  *NOTE: If there is a shortage of pegylated liposomal doxorubicin hydrochloride, patients receive epirubicin hydrochloride IV over 15-20 minutes on day 1.
  Interventions: Drug: pegylated liposomal doxorubicin hydrochloride; Drug: epirubicin hydrochloride; Drug: carboplatin; Procedure: therapeutic conventional surgery; Drug: paclitaxel; Other: laboratory biomarker analysis; Other: quality-of-life assessment

INTERVENTIONS:
Drug: pegylated liposomal doxorubicin hydrochloride — Given IV
  Other Names: CAELYX; Dox-SL; DOXIL; doxorubicin hydrochloride liposome; LipoDox
Drug: epirubicin hydrochloride — Given IV
  Other Names: 4'-epi-doxorubicin HCl; 4'-epiadriamycin
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Procedure: therapeutic conventional surgery — Undergo definitive surgery
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Other: laboratory biomarker analysis — Correlative studies
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This phase II trial studies how well pegylated liposomal doxorubicin hydrochloride and carboplatin followed by surgery and paclitaxel work in treating patients with stage II-III breast cancer that does not have estrogen receptors, progesterone receptors, or large amounts of human epidermal growth factor receptor 2 (HER2)/neu protein (triple negative). Drugs used in chemotherapy, such as pegylated liposomal doxorubicin hydrochloride, carboplatin, and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving pegylated liposomal doxorubicin hydrochloride and carboplatin before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving pegylated liposomal doxorubicin hydrochloride and carboplatin followed by surgery and paclitaxel may be an effective treatment for breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the rate of pathologic complete response with treatment of liposomal doxorubicin (pegylated liposomal doxorubicin hydrochloride) and carboplatin in patients with estrogen receptor (ER), progesterone receptor (PR), HER2 negative breast cancer (triple negative breast cancer [TNBC]).

SECONDARY OBJECTIVES:

I. To determine the recurrence free survival (RFS), 2-year RFS, and overall survival (OS) after treatment with neoadjuvant liposomal doxorubicin and carboplatin followed by definitive breast surgery and then weekly paclitaxel in patients with ER, progesterone receptor (PgR), HER2 negative breast cancer.

II. To describe the mutational spectrum of tumors found in primary, untreated ER, PgR, HER2 negative breast cancer and their association with pathologic complete response to neoadjuvant pegylated liposomal doxorubicin hydrochloride (doxil) and carboplatin.

III. To determine functional significance of genomic landscape in predicting drug response using patient derived xenograft (PDX) and ex vivo models.

OUTLINE:

NEOADJUVANT: Patients receive pegylated liposomal doxorubicin hydrochloride* intravenously (IV) over 90 minutes and carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.

ADJUVANT: Patients undergo definitive surgery at the discretion of the treating physician. Patients then receive paclitaxel IV over 60 minutes once weekly for 12 weeks in the absence of disease progression or unacceptable toxicity.

*NOTE: If there is a shortage of pegylated liposomal doxorubicin hydrochloride, patients receive epirubicin hydrochloride IV over 15-20 minutes on day 1.

After completion of study treatment, patients are followed up every 6 months for up to 20 years.

ELIGIBILITY:
Inclusion Criteria:

* Women with previously untreated, unilateral stage II-III breast cancer, ER/PgR/HER2 negative (ER =< 5%, PgR =< 5%, HER2 0-1+ by immunohistochemistry [IHC] or fluorescence in situ hybridization [FISH] =< 2.0); if clinically negative lymph nodes, tumor size should be minimum 1.0 cm and identifiable under office-based ultrasound guidance
* Negative serum or urine beta-human chorionic gonadotropin (hCG) pregnancy test at screening for patients of child-bearing potential within one week prior to enrollment
* Patients with reproductive potential must use an adequate contraceptive method (e.g. abstinence, intrauterine device, oral contraceptives, barrier device with spermicide or surgical sterilization) during treatment and for three months after completing treatment
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status < 2
* Life expectancy >= 52 weeks excluding their diagnosis of breast cancer
* Absolute neutrophil count (ANC) >= 1,500 cells/mm^3
* Platelets >= 100,000 cells/mm^3
* Hemoglobin > 9.0 g/dL
* Creatinine < 2.5 mg/dL
* Total bilirubin < 1.5 X upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2.5 X institutional ULN
* Patients must have normal cardiac function, as evidenced by a left ventricular ejection fraction (LVEF) within institutional normal limits; echocardiogram may be used if multi gated acquisition (MUGA) scan is not available, but the same test must be used throughout the study to evaluate LVEF
* Computed tomography of the chest, abdomen, and pelvis (CT CAP) and bone scan performed within 30 days prior to study entry and does not demonstrate metastatic disease
* Patients may not receive concurrent treatment with other investigational or commercial agent(s) for treatment of their breast cancer
* The patient or, if applicable, her legally authorized representative must have signed and dated an Institutional Review Board (IRB)-approved consent form that conforms to federal and institutional guidelines
* Patients must be eligible to undergo surgery, either lumpectomy or mastectomy for local treatment of the breast cancer; surgical margins at discretion of surgeon per National Comprehensive Cancer Network (NCCN) guidelines; axillary exploration at discretion of surgeon but all patients minimally have sentinel lymph node evaluation at time of surgery
* Imaging by magnetic resonance imaging (MRI), ultrasound and/or mammogram and physical exam to document lesions size must be performed within 30 days of study entry
* Must not exhibit a non-healing wound or any skin breakdown
* Before administering liposomal doxorubicin, patients must wait 4-6 weeks after surgery
* Submission of tumor samples from the diagnostic biopsy and breast surgery is required for all patients

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Second primary malignancy except most situ carcinoma (e.g. in situ carcinoma of the cervix, adequately treated non-melanomatous carcinoma of the skin) or other malignancy treated at least 5 years previously with no evidence of recurrence
* Definitive clinical or radiologic evidence of metastatic disease; imaging must have been performed no greater than 30 days prior to initiation of chemotherapy
* Diagnosis of inflammatory breast cancer
* History of hypersensitivity reactions attributed to a conventional formulation of doxorubicin hydrochloride (HCL) or the components of doxil, paclitaxel, or carboplatin
* Serious concomitant systemic disorders (including active infections or chronic infection requiring suppressive antibiotics) that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator
* Myocardial infarct or unstable angina within 6 months before enrollment, New York Heart Association (NYHA) class II or greater heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, clinically significant pericardial disease, valvular disease with documented compromise in cardiac function, or electrocardiographic evidence of acute ischemic or active conduction system abnormalities
* Prior anthracycline, platinum salt, or taxane for any malignancy
* Known or active hepatitis B or C with abnormal liver function tests
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Intrinsic lung disease resulting in moderate to severe dyspnea
* History of a major organ allograft or condition requiring chronic immunosuppression, e.g., kidney, liver, lung, heart, bone marrow transplant, or autoimmune diseases; this includes treatment with corticosteroids within one month (dose of >= 10 mg/day methylprednisolone equivalent) (excluding inhaled steroids); patients who have received corneal transplants, cadaver skin, or bone transplants are eligible
* Nervous system disorder (paresthesias, peripheral motor neuropathy, or peripheral sensory neuropathy) >= grade 2, per the Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0)
* Conditions that would prohibit administration of corticosteroids

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-02-25 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2041-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Hirshfield, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 62 participants were enrolled, nine participants withdrew consent either prior to treatment or completion of neoadjuvant therapy and or surgery.
Groups:
- Treatment (Doxil, Carboplatin, Surgery, Paclitaxel): Participants received 4 cycles of neoadjuvant Lipposomal doxorubicin (DOX)+Carboplatin(CAR) administered every 28 days, followed by definitive breast surgery and adjuvant paclitaxel 80 mg/m2 administered weekly
Period: Overall Study
Arm/Group | Treatment (Doxil, Carboplatin, Surgery, Paclitaxel)
Started | 62
Completed | 53
Not Completed | 9
Not completed — Withdrew consent | 9

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Doxil, Carboplatin, Surgery, Paclitaxel): NEOADJUVANT: Patients receive pegylated liposomal doxorubicin hydrochloride* IV over 90 minutes and carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  ADJUVANT: Patients undergo definitive surgery at the discretion of the treating physician. Patients then receive paclitaxel IV over 60 minutes once weekly for 12 weeks in the absence of disease progression or unacceptable toxicity.
  *NOTE: If there is a shortage of pegylated liposomal doxorubicin hydrochloride, patients receive epirubicin hydrochloride IV over 15-20 minutes on day 1.
  pegylated liposomal doxorubicin hydrochloride: Given IV
  epirubicin hydrochloride: Given IV
  carboplatin: Given IV
  therapeutic conventional surgery: Undergo definitive surgery
  paclitaxel: Given IV
  laboratory biomarker analysis: Correlative studies
  quality-of-life assessment: Ancillary studies
Arm/Group | Treatment (Doxil, Carboplatin, Surgery, Paclitaxel)
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 13
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 53

OUTCOME MEASURES:

1. Primary Outcome: Rate of Pathologic Complete Response (pCR) Based on Response Evaluation Criteria in Solid Tumors Criteria
Description: The pCR rate will first be determined as proportions and calculating its 95% confidence interval. To study the association between pCR response (yes/no) and the presence of gross residual disease, type and number of mutations, clinical lymph node status (positive/negative), tumor size (< 2 cm/>= 2 cm) based on p53, logistic regression analysis will be used, controlling for cancer treatment and disease stage and other covariates if numbers allow.
Time Frame: Disease was evaluated at baseline to after four cycles every 28 days and then after twelve weeks of treatment after surgery (up to 28 weeks from baseline).
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (Doxil, Carboplatin, Surgery, Paclitaxel): Participants received 4 cycles of neoadjuvant liposomal doxorubicin (DOX)+carboplatin (CAR) administered every 28 days, followed by definitive breast surgery and adjuvant paclitaxel 80 mg/m2 administered weekly.
Arm/Group | Treatment (Doxil, Carboplatin, Surgery, Paclitaxel)
Number analyzed (Participants) | 53
Participants | 16

2. Secondary Outcome: OS
Description: Survival functions will be computed using the Kaplan-Meier method, and compared between mutation status using the log-rank test. Adjustment for additional covariates, such as cancer treatment and disease stage, will be performed using Cox proportional hazards regression analysis if numbers allow.
Time Frame: Time from initiation of chemotherapy until death from any cause, assessed up to 20 years
Reporting Status: Not Posted, anticipated posting 2041-07

3. Secondary Outcome: Mutational Spectrum of Tumors
Description: The Cox model analysis will be used to study the association between cancer recurrence and the presence of specific mutations with IHC parameters, e.g. p53, Ki67, apoptotic markers (cleaved caspase 3), phosphorylated proteins in targeted pathways, gamma-H2A histone family, member X for deoxyribonucleic acid damage. All test procedures will be done at significance level 5%. It will be determined which tumors with gross residual disease are sensitive to targeted agent, cytotoxins, or the combination as a function of mutational profile and will be tested for additive and synergistic effects.
Time Frame: Time from initiation of chemotherapy until death from any cause, assessed up to 20 yearsUp to 20 years
Reporting Status: Not Posted, anticipated posting 2041-07

ADVERSE EVENTS:
Time Frame: Disease was evaluated at baseline to after four cycles every 28 days and then after twelve weeks of treatment after surgery (up to 28 weeks from baseline).
Groups:
- Treatment (Doxil, Carboplatin, Surgery, Paclitaxel): Participants received 4 cycles of neoadjuvant DOX+CAR administered every 28 days, followed by definitive breast surgery and adjuvant paclitaxel 80 mg/m2 administered weekly.
Arm/Group | Treatment (Doxil, Carboplatin, Surgery, Paclitaxel)
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 22/53
Other Adverse Events (participants affected / at risk) | 53/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Doxil, Carboplatin, Surgery, Paclitaxel) (N=53)
febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 16 (20)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3)
Pruritis (Gastrointestinal disorders) | 1 (5)
Mucositis (Infections and infestations) | 2 (7)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Doxil, Carboplatin, Surgery, Paclitaxel) (N=53)
Fatigue (General disorders) | 50 (79)
Anemia (Blood and lymphatic system disorders) | 44 (110)
Alopecia (General disorders) | 10 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/96/NCT02315196/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/96/NCT02315196/SAP_001.pdf
  • Informed Consent Form (2015-07-31): https://cdn.clinicaltrials.gov/large-docs/96/NCT02315196/ICF_002.pdf